CLINICAL TRIAL: NCT00646919
Title: Double-Blind Prospective Study Concerning the Connection Between Positive Nasal Culture for Staphyloccoci in Pediatric Patients Undergoing Any Elective Surgery in the Out-Patient Clinic in the Hillel Yaffe Medical Center, Over a Period of One Year
Brief Title: Preoperative Nasal Swabs From Pediatric Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Other Study IDs: HY56/2007
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Staphylococcal Infections
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: All pre-operative pediatric patients in our outpatient clinic
  Interventions: Procedure: Nose swab

INTERVENTIONS:
Procedure: Nose swab

SUMMARY:
We intend to take a nasal swab from each pediatric pre-operative patient in our out-clinic with the intention of looking for a connection between positive operative incisions and a positive nasal swab. The patients will be in the out-patient clinic for a few hours, and will be examined post-operatively after one week. Those with positive nasal swabs will be advised to apply a nasal cream (Mupirocin)in their noses for one week. Our hypothesis is that there is a correlation between positive nasal swabs and positive incision infections.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients attending outpatient surgery clinic

Exclusion Criteria:

* All others

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pediatric patients attending our outpatient surgery clinic
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel